CLINICAL TRIAL: NCT03085758
Title: A Double-Blind, Placebo-Controlled, Randomized, Multicenter, Proof of Concept and Dose-Finding Phase II Clinical Trial to Investigate the Safety, Tolerability and Efficacy of ADRECIZUMAB in Patients With Septic Shock and Elevated Adrenomedullin
Brief Title: Treatment of Patients With Early Septic Shock and Bio-Adrenomedullin(ADM) Concentration > 70 pg/ml With ADRECIZUMAB
Acronym: AdrenOSS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adrenomed AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADR-02
Record Dates: First submitted 2017-02-22; First posted 2017-03-21 (Actual); Results first posted 2021-03-24 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-01

CONDITIONS: Septic Shock
Keywords: Early Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — enibarcimab

STUDY DESIGN:
Intervention Model Description: Double Blind, Placebo-Controlled, Randomized, Multicenter Proof of Concept and Dose-Finding Phase II Clinical Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Arm A (Experimental): Intravenous infusion over approximately 1 hour of single i.v. dose of 2 mg/kg Adrecizumab (treatment arm A)
  Interventions: Biological: Adrecizumab
- Treatment Arm B (Experimental): Intravenous infusion over approximately 1 hour of single i.v. dose of 4 mg/kg Adrecizumab (treatment arm B)
  Interventions: Biological: Adrecizumab
- Control group (Placebo Comparator): Intravenous infusion over approximately 1 hour of single i.v. dose of Placebo of Adrecizumab (control group)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Adrecizumab — Single i.v. dose of 2 mg/kg (treatment arm A) or 4 mg/kg (treatment arm B)
  Arms: Treatment Arm A; Treatment Arm B
Biological: Placebo — Single i.v. dose of placebo (control group)
  Arms: Control group

SUMMARY:
This is a double-blind, placebo-controlled, randomized, multicenter proof of concept and dose-finding phase II study using two doses of ADRECIZUMAB in patients with early septic shock and a bio-ADM plasma concentration at admission of > 70 pg/ml.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, multicenter proof of concept and dose-finding phase II study using two doses of ADRECIZUMAB in patients with early septic shock and a bio-ADM plasma concentration at admission of > 70 pg/ml.

"Early" septic shock is defined as a life-threatening organ dysfunction due to dysregulated host response to a proven or suspected infection which leads to a decline of Mean Arterial Pressure (MAP) < 65 mmHg, which is refractory to fluid resuscitation and requires vasopressors. Early is defined as a maximum of less than 12 hours between onset of the cardiovascular organ-dysfunction and administration of ADRECIZUMAB. Refractoriness to fluid resuscitation is defined as a lack of response to the administration of 30 mL of fluid per kilogram of body weight or is determined according to a clinician's assessment of inadequate hemodynamic results.

It is intended to enroll 300 patients from surgical, medical and mixed ICU at multiple centers in Europe.

All patients will be treated according to "International Guidelines for Management of Severe Sepsis and Septic Shock".

Eligible patients (confirmed by central verification) will be randomized (1:1:2) to ADRECIZUMAB treatment arm A (2 mg/kg) or to ADRECIZUMAB treatment arm B (4 mg/kg) or to placebo as control group. Patients assigned to the treatment arm A or B will be administered a single dose of ADRECIZUMAB as intravenous infusion over approximately 1 hour; patients assigned to the control group will be administered placebo as intravenous infusion over approximately 1 hour.

As long as the patients are on the ICU, daily measurements of clinical signs and laboratory data will be collected for safety reasons and for determination of Sequential Organ Failure Assessment Score (SOFA score). Additional blood samples for central laboratory analyses will be taken at inclusion on day 1, day 3, day 5, day 7 or day of discharge (whatever comes first) for measurement of biomarkers.

The SOFA score and its components will be determined daily for all patients over the entire stay on the ICU (28 days or until discharge whatever comes first). Safety monitoring for each patient will begin at the time of signing the Informed Consent Form and continue for 90 days after end of short-term infusion of study medication.

At selected study centers a pharmacokinetic (PK) substudy will be performed to determine the profile of ADRECIZUMAB in 80 randomized patients.

An interim analysis for efficacy is planned after 50% of patients have completed the study (n=150).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by patient or legal representative (according to country - specific regulations)
2. Male and female patient, age ≥ 18 years
3. Body weight 50 kg - 120 kg
4. Bio-ADM concentration > 70 pg/ml
5. Patient with early septic shock (start of vasopressor therapy < 12 hours)
6. Women of childbearing potential must have a negative serum or urine pregnancy test before randomization
7. Highly effective method of contraception must be maintained for 6 months after study start by women of childbearing potential and sexually active men.
8. No care limitation

Exclusion Criteria:

1. Moribund
2. Pre-existing unstable condition (e.g. a recent cerebral hemorrhage or infarct, a recent acute unstable myocardial infarction (all < 3 months), congestive heart failure - New York Heart Association (NYHA) Class IV
3. Patients that required cardiopulmonary resuscitation in the last 4 weeks prior to evaluation for enrollment
4. Severe Chronic Obstructive Pulmonary Disease (COPD) with chronic oxygen need at home (GOLD IV)
5. Any organ or bone marrow transplant within the past 24 weeks
6. Uncontrolled serious hemorrhage (≥ 2 units of blood / platelets in the previous 24 hrs.). Patients may be considered for enrollment if bleeding has stopped and patient is otherwise qualified
7. Uncontrolled hematological / oncological malignancies
8. Absolute neutropenia < 500 per µL
9. Severe chronic liver disease (Child-Pugh C)
10. Systemic fungal infection or active tuberculosis
11. Neuromuscular disorders that impact breathing / spontaneous ventilation
12. Burns > 30% of body surface
13. Plasmapheresis
14. Breastfeeding women
15. Participation in a clinical trial involving another investigational drug within 4 weeks prior to inclusion
16. Unwilling or unable to be fully evaluated for all follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Zimmermann, Dr., Study Director — Adrenomed AG
Locations (30):
- Belgium (4):
  - Clinique Universitaire Saint-Luc (UCL Bruxelles), Brussels
  - Antwerp University Hospital (UZA), Critical Care Medicine, Edegem
  - Groupe Jolimont, Hospitalier de Jolimont, Haine-Saint-Paul
  - Clinique St. Pierre, Intensive Care, Ottignies
- France (16):
  - Medical Intensive Care Medicine, Centre hospital - universitaire, Angers, Cedex
  - CH Victor Dupouy, Argenteuil, Cedex
  - Hopital Beaujon; Anesthesie Reanimation, Clichy, Cedex
  - CHU de Limoges, Limoges, Cedex
  - CHU de Nantes; Medicine Intensive Reanimation, Nantes, Cedex
  - CHRU Bretonneau, Medecine Intensive Réanimation, Tours, Cedex
  - University Hospital of Clermont-Ferrand, Dept. of Perioperative Medicine, Clermont-Ferrand
  - AP-HP, Hopital Louis Mourier, Réanimation Médicale, Colombes
  - CHD-Vendée, La Roche-sur-Yon
  - Hôpital de Bicêtre, Service d'anesthésie-réanimation chirurgicale, Le Kremlin-Bicêtre
  - Hôpital Lariboisière, Dept. d'Anesthesie, Paris
  - Hôpital Lariboisière, Réanimation Médicale et Traumatologique, Paris
  - Hôpital Saint-Louis, Service d'Anesthésie-Réanimation, Paris
  - Hôpital Européen Georges Pompidou, Service d'Anesthésie-Réanimation Chirurgicale, Université Paris Descartes, Paris
  - Nouvel Hopital Civil, Strasbourg
  - Hôpital de Hautepierre , Hôpitaux Universitaires de Strasbourg, Unité de Réanimation Chirurgicale, Service d'Anesthésie-Réanimation Chirurgicale, Strasbourg
- Germany (5):
  - Universitätsklinikum Aachen, Klinik für Operative Intensivmedizin, Aachen
  - Universitätsklinikum Hamburg-Eppendorf Klinik für Intensivmedizin, Hamburg
  - Universitätsklinikum Jena Klinik für Anästhesiologie und Intensivmedizin, Jena
  - Universitätsklinikum Münster Klinik für Anästhesiologie, operative Intensivmedizin und Schmerztherapie, Münster
  - Universitätsmedizin Rostock Klinik und Poliklinik für Anästhesiologie und Intensivtherapie, Rostock
- Netherlands (5):
  - Gelderse Vallei Hospital, Department of Intensive Care, Ede
  - Medisch Spectrum Twente, Department of Intensive Care, Enschede
  - Zuyderland Medical Center, Department of Intensive Care, Heerlen
  - Radboud UMC Intensive Care, Nijmegen
  - Canisius-Wilhelmina-Ziekenhuis (CWZ), Intensive Care, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laterre PF, Pickkers P, Marx G, Wittebole X, Meziani F, Dugernier T, Huberlant V, Schuerholz T, Francois B, Lascarrou JB, Beishuizen A, Oueslati H, Contou D, Hoiting O, Lacherade JC, Chousterman B, Pottecher J, Bauer M, Godet T, Karakas M, Helms J, Bergmann A, Zimmermann J, Richter K, Hartmann O, Pars M, Mebazaa A; AdrenOSS-2 study participants. Safety and tolerability of non-neutralizing adrenomedullin antibody adrecizumab (HAM8101) in septic shock patients: the AdrenOSS-2 phase 2a biomarker-guided trial. Intensive Care Med. 2021 Nov;47(11):1284-1294. doi: 10.1007/s00134-021-06537-5. Epub 2021 Oct 4. PMID 34605947
- [Derived] Geven C, Blet A, Kox M, Hartmann O, Scigalla P, Zimmermann J, Marx G, Laterre PF, Mebazaa A, Pickkers P. A double-blind, placebo-controlled, randomised, multicentre, proof-of-concept and dose-finding phase II clinical trial to investigate the safety, tolerability and efficacy of adrecizumab in patients with septic shock and elevated adrenomedullin concentration (AdrenOSS-2). BMJ Open. 2019 Feb 19;9(2):e024475. doi: 10.1136/bmjopen-2018-024475. PMID 30782906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 08-Dec-2017 Last patient completed: 20-Dec-2019 Total study duration: 25 months
Groups:
- Treatment Arm A: Intravenous infusion over approximately 1 hour of single i.v. dose of 2 mg/kg Adrecizumab
  Adrecizumab: Single i.v. dose of 2 mg/kg
- Treatment Arm B: Intravenous infusion over approximately 1 hour of single i.v. dose of 4 mg/kg Adrecizumab
  Adrecizumab: Single i.v. dose of 4 mg/kg
- Control Group: Intravenous infusion over approximately 1 hour of single i.v. dose of Placebo of Adrecizumab
  Placebo: Single i.v. dose of placebo
Period: Overall Study
Arm/Group | Treatment Arm A | Treatment Arm B | Control Group
Started | 72 | 77 | 152
Completed | 43 | 49 | 96
Not Completed | 29 | 28 | 56
Not completed — Death | 26 | 24 | 53
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Refusal to recall it up to day 90 | 0 | 0 | 1
Not completed — Pt seen by doctor in digestive surgery | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Control Group | Total
Number analyzed (Participants) | 72 | 77 | 152 | 301
Age, Continuous [Mean (Full Range); unit: years] | 66.2 [30 to 94] | 68.8 [18 to 89] | 69.3 [21 to 94] | 68.4 [18 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 66 | 117
  Male | 45 | 53 | 86 | 184
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 3 | 5
  Black | 1 | 1 | 0 | 2
  Caucasian | 56 | 58 | 107 | 221
  Other | 1 | 0 | 1 | 2
  Not reported | 13 | 17 | 41 | 71
Region of Enrollment [Number; unit: participants]
  Netherlands | 8 | 10 | 19 | 37
  Belgium | 23 | 24 | 43 | 90
  France | 30 | 30 | 64 | 124
  Germany | 11 | 13 | 26 | 50
Location before ICU admission [Number; unit: participants]
  Home | 7 | 9 | 8 | 24
  Hospital | 65 | 68 | 144 | 277
Origin of sepsis [Number; unit: participants]
  Peritonitis | 12 | 17 | 36 | 65
  Lung | 14 | 17 | 32 | 63
  Urinary tract | 18 | 10 | 26 | 54
  Skin and soft tissue | 2 | 8 | 14 | 24
  Bile duct infection | 4 | 5 | 6 | 15
  Blood stream | 4 | 5 | 6 | 15
  Central nervous system | 1 | 1 | 1 | 3
  Catheter | 0 | 0 | 4 | 4
  Other | 17 | 14 | 27 | 58
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — Population: Treatment group A Row population differs from the Overall because height was not determined for one subject, therefore, no BMI was calculated.
  Treatment group C Row population differs from the Overall because height was not determined for one subject, therefore, no BMI was calculated.
  kg/m^2
    number analyzed (Participants) | 71 | 77 | 151 | 299
    (all) | 26.41 [16.7 to 45.7] | 26.72 [17.0 to 43.3] | 27.78 [14.1 to 45.5] | 27.18 [14.1 to 45.7]
Body temperature [Mean (Full Range); unit: degrees C] — Population: Treatment group A Row population differs from the Overall because body temperature was not done for 6 subjects.
  Treatment group B Row population differs from the Overall because body temperature was not done for 4 subjects.
  Treatment group C Row population differs from the Overall because body temperature was not done for 7 subjects.
  degrees C
    number analyzed (Participants) | 66 | 73 | 145 | 284
    (all) | 37.06 [34.6 to 39.9] | 36.97 [33.4 to 39.9] | 37.08 [33.8 to 40.5] | 37.05 [33.4 to 40.5]
Heart rate [Mean (Full Range); unit: bpm] | 104.38 [51.0 to 158.0] | 97.40 [60.0 to 151.0] | 96.37 [44.0 to 153.0] | 98.55 [44.0 to 158.0]
Mean arterial pressure [Mean (Full Range); unit: mmHg] | 73.18 [43.0 to 99.0] | 71.35 [32.0 to 104.0] | 72.49 [22.0 to 110.0] | 72.36 [22.0 to 110.0]
Respiratory rate [Mean (Full Range); unit: breaths/min] — Population: Treatment group A Row population differs from the Overall because respiratory rate was not done for 2 subjects
  Treatment group C Row population differs from the Overall because respiratory rate was not done for 3 subjects
  breaths/min
    number analyzed (Participants) | 70 | 77 | 149 | 296
    (all) | 23.63 [8.0 to 44.0] | 21.90 [10.0 to 37.0] | 21.96 [8.0 to 36.0] | 22.34 [8.0 to 44.0]
Bio-ADM [Mean (Full Range); unit: pg/mL (local)] — bio-ADM measures the plasma level of the biological active Adrenomedullin, a vasoactive hormone that regulates blood pressure and vascular integrity
  Note results characterized as "3000" are to be read as >3000
  pg/mL (local) | 284.30 [74.9 to 1967.1] | 305.15 [74.6 to 2328.9] | 755.92 [74.3 to 3000] | 527.80 [74.3 to 3000]
Blood lactate [Mean (Full Range); unit: mmol/L] — Population: Treatment group A Row population differs from the Overall because blood lactate was not done for 4 subjects Treatment group B Row population differs from the Overall because blood lactate was not done for 2 subjects Treatment group C Row population differs from the Overall because blood lactate was not done for 3 subjects
  mmol/L
    number analyzed (Participants) | 68 | 75 | 149 | 292
    (all) | 4.11 [0.8 to 15.0] | 4.19 [0.9 to 17.0] | 4.23 [0.6 to 64.0] | 4.19 [0.6 to 64.0]
Creatinine [Mean (Full Range); unit: μmol/L] — Population: Treatment group A Row population differs from the Overall because creatinine was not done for 1 subject Treatment group B Row population differs from the Overall because creatinine was not done for 1 subject
  μmol/L
    number analyzed (Participants) | 71 | 76 | 152 | 299
    (all) | 189.649 [31.82 to 582.00] | 199.891 [53.04 to 834.50] | 192.801 [32.10 to 912.29] | 193.854 [31.82 to 912.29]
Apache II Score [Mean (Full Range); unit: units on a scale] — Minimum score = 0; maximum score = 71. Increasing score is associated with increasing risk of hospital death. Population: Treatment group A Row population differs from the Overall because Apache II Score was not done for 10 subjects Treatment group B Row population differs from the Overall because Apache II Score was not done for 11 subjects Treatment group C Row population differs from the Overall because Apache II Score was not done for 8 subjects
  units on a scale
    number analyzed (Participants) | 62 | 66 | 144 | 272
    (all) | 31.4 [17 to 42] | 31.8 [20 to 42] | 31.5 [14 to 53] | 31.6 [14 to 53]
Sequential Organ Failure Assessment (SOFA) Score [Mean (Full Range); unit: units on a scale] — The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems.
  SOFA score: Minimum possible score is 0, maximum is 24. A higher score meas a worse outcome. Population: Treatment group A Row population differs from the Overall because SOFA Score was not done for 11 subjects Treatment group B Row population differs from the Overall because SOFA Score was not done for 16 subjects Treatment group C Row population differs from the Overall because SOFA Score was not done for 20 subjects
  units on a scale
    number analyzed (Participants) | 61 | 61 | 132 | 254
    (all) | 10.1 [4 to 17] | 10.0 [5 to 16] | 9.6 [4 to 16] | 9.9 [4 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Endpoints for Primary Objective (Safety and Tolerability of Adrecizumab: Mortality)
Description: The endpoints for the primary objective is mortality evaluated over the 90 days study period.
Time Frame: 90 days
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: days
Groups:
- Adrecizumab Overall: Treatment Arm A and Treatment Arm B combined
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
days | 63.1453 (4.0940) | 63.1578 (3.5967) | 64.5744 (2.7582) | 63.9809 (2.9466)

2. Primary Outcome: Endpoints for Primary Objective (Safety and Tolerability of Adrecizumab: Interruption of Infusion)
Description: The endpoints for the primary objective are to determine over the 90 days study period: Interruption of infusion due to intolerability of ADRECIZUMAB
Time Frame: 90 days
Population: Safety Analysis Set
Measure: Number; unit: Interruptions
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
Interruptions | 0 | 1 | 1 | 0

3. Primary Outcome: Endpoints for Primary Objective (Safety and Tolerability of Adrecizumab: Frequency of TEAEs)
Description: The endpoints for the primary objective are to determine over the 90 days study period. Number of participants with treatment-emergent adverse events per treatment group.
Time Frame: 90 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
Participants | 68 | 74 | 142 | 142

4. Primary Outcome: Endpoints for Primary Objective (Safety and Tolerability of Adrecizumab: Severity and Frequency of TEAEs) - Mild Severity
Description: The endpoints for the primary objective are to determine over the 90 days study period. Number of participants with treatment-emergent adverse events per treatment group with mild severity treatment emergent events.
Time Frame: 90 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
Participants | 39 | 46 | 85 | 82

5. Primary Outcome: Endpoints for Primary Objective (Safety and Tolerability of Adrecizumab: Severity and Frequency of TEAEs) - Moderate Severity
Description: The endpoints for the primary objective are to determine over the 90 days study period. Number of participants with treatment-emergent adverse events per treatment group with moderate severity treatment emergent events.
Time Frame: 90 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
Participants | 54 | 60 | 114 | 109

6. Primary Outcome: Endpoints for Primary Objective (Safety and Tolerability of Adrecizumab: Severity and Frequency of TEAEs) - Severe Severity
Description: The endpoints for the primary objective are to determine over the 90 days study period. Number of participants with treatment-emergent adverse events per treatment group with severe severity treatment emergent events.
Time Frame: 90 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
Participants | 51 | 54 | 105 | 108

7. Secondary Outcome: Efficacy to be Determined by Sepsis Support Index (SSI)
Description: The primary efficacy endpoint of this study is the Sepsis Support Index (SSI) defined as: days with organ support or dead within 14 day follow up More precisely: In the time frame of 14 day follow-up, each day on support with vasopressor, and/or mechanical ventilation, and/or renal dysfunction (defined as renal SOFA = 4), or not alive, is counted as 1. The sum over the follow up period is defined as SSI.
  Minimum value possible is 0, maximum value is 14. A higher score means a worse outcome.
Time Frame: 14 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 71 | 75 | 146 | 151
score on a scale | 8.4 (5.16) | 9.1 (5.20) | 8.8 (5.18) | 8.1 (5.41)

8. Secondary Outcome: Sepsis Support Index (SSI)
Description: Sepsis Support Index (SSI) at 28 day follow-up Minimum value possible is 0, maximum value is 14. A higher score means a worse outcome.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 70 | 75 | 145 | 151
score on a scale | 13.3 (10.91) | 14.6 (10.76) | 14.0 (10.82) | 12.8 (11.14)

9. Secondary Outcome: Penalized Sepsis Support Index (pSSI) at 14 Day Follow-up
Description: Penalized Sepsis Support Index (pSSI) at day 14, defined similar to the SSI with the exception that patients that die get penalized by assigning the maximum value, i.e. the pSSI is set to 14 or 28, respectively.
  Minimum value possible is 0, maximum value is 14. A higher score means a worse outcome.
Time Frame: day 14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 71 | 75 | 146 | 151
score on a scale | 8.5 (5.26) | 9.1 (5.20) | 8.8 (5.22) | 8.1 (5.42)

10. Secondary Outcome: Persistent Organ Dysfunction or Death at 14 and 28 Day Follow-up
Description: Persistent organ dysfunction or death at 14 and 28 day follow-up. Count of participants with either persistent organ dysfunction or death at Day 14 and Day 28. Persistent Organ Dysfunction is defined as the persistence of organ dysfunction requiring supportive technologies during the convalescent phase of critical illness and it is present when a patient has an ongoing requirement for vasopressors, dialysis, or mechanical ventilation at the outcome assessments time points, as defined by Heyland et al.; Persistent organ dysfunction plus death: a novel,composite outcome measure for critical care trials. Critical Care 2011, 15.
Time Frame: day 14 and day 28
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
Participants
  Day 14 | 29 | 37 | 66 | 63
  Day 28 | 25 | 25 | 50 | 49

11. Secondary Outcome: Mortality Rate
Description: Day 28 mortality rate
Time Frame: day 28
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: days
Groups:
- Adrecizumab Overall: Treatment Group A and Treatment Group B combined
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
days | 20.3484 (0.8694) | 17.5630 (0.6592) | 20.5162 (0.5903) | 22.8783 (0.7627)

12. Secondary Outcome: SSI and pSSI Excluding the Renal Component
Description: Sepsis Support Index (SSI) and penalized Sepsis Support Index (pSSI) excluding the renal component. pSSI is a version of the SSI where mortality is given extra weight: Patients being alive during the 14 days' follow up will have an SSI ranging up to 14, while patients who died within that period will be assigned a score of "14 plus the number of days not being alive". Thus the SSI and pSSI score may range between zero and 28. A higher score means a worse outcome. The number of participants analyzed differs per row due to missing data.
Time Frame: day 14 and day 28
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 146 | 152
score on a scale
  SSI Day 14: number analyzed (Participants) | 71 | 75 | 146 | 151
  SSI Day 14 | 8.0 (5.21) | 9.0 (5.24) | 8.5 (5.24) | 7.9 (5.42)
  SSI Day 28: number analyzed (Participants) | 71 | 75 | 146 | 151
  SSI Day 28 | 12.9 (11.03) | 14.3 (10.80) | 13.6 (10.90) | 12.6 (11.17)
  pSSI Day 14: number analyzed (Participants) | 71 | 75 | 146 | 151
  pSSI Day 14 | 8.1 (5.32) | 9.0 (5.24) | 8.6 (5.28) | 7.9 (5.43)
  pSSI Day 28: number analyzed (Participants) | 71 | 75 | 146 | 151
  pSSI Day 28 | 13.4 (11.47) | 14.5 (10.92) | 14.0 (11.17) | 12.9 (11.39)

13. Secondary Outcome: SSI Weighted for Mortality
Description: Sepsis Support Index (SSI) Weighted for Mortality. Minimum value possible is 0, maximum value is 14. A higher score means a worse outcome.
Time Frame: day 14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 71 | 75 | 146 | 150
score on a scale | 10.2 (7.76) | 10.7 (7.65) | 10.5 (7.68) | 9.9 (8.41)

14. Secondary Outcome: Individual Sepsis Support Index Components
Description: Individual Sepsis Support Index (SSI) components (hemodynamic, respiratory and renal failure) with and without mortality.
  Minimum value possible is 0, maximum value is 14. A higher score means a worse outcome. The number of participants analyzed differs per row due to missing data.
Time Frame: day 14 and day 28
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
score on a scale
  SSI cardiac component day 14: number analyzed (Participants) | 57 | 64 | 121 | 119
  SSI cardiac component day 14 | 4.0 (2.95) | 5.4 (4.01) | 4.7 (3.60) | 4.6 (3.84)
  SSI cardiac component day 28: number analyzed (Participants) | 53 | 58 | 111 | 109
  SSI cardiac component day 28 | 4.8 (5.03) | 5.8 (5.61) | 5.3 (5.35) | 4.7 (4.55)
  SSI respiratory component day 14: number analyzed (Participants) | 57 | 64 | 121 | 119
  SSI respiratory component day 14 | 5.4 (5.41) | 7.3 (5.98) | 6.4 (5.78) | 5.1 (5.57)
  SSI respiratory component day 28: number analyzed (Participants) | 53 | 58 | 111 | 109
  SSI respiratory component day 28 | 6.9 (9.14) | 9.6 (9.85) | 8.3 (9.57) | 5.8 (8.08)
  SSI renal failure component day 14: number analyzed (Participants) | 57 | 64 | 121 | 119
  SSI renal failure component day 14 | 1.3 (3.55) | 1.5 (3.27) | 1.4 (3.39) | 1.4 (3.37)
  SSI renal failure component day 28: number analyzed (Participants) | 52 | 58 | 110 | 107
  SSI renal failure component day 28 | 1.9 (5.30) | 1.9 (4.63) | 1.9 (4.93) | 1.4 (3.79)
  SSI death component day 14: number analyzed (Participants) | 71 | 75 | 146 | 151
  SSI death component day 14 | 1.7 (3.86) | 1.6 (4.02) | 1.6 (3.93) | 2.0 (4.34)
  SSI death component day 28: number analyzed (Participants) | 71 | 75 | 146 | 151
  SSI death component day 28 | 4.9 (9.23) | 4.5 (9.07) | 4.7 (9.12) | 5.5 (9.81)

15. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Score : Composite Measure: SOFA Score and Its Changes Over Time
Description: Sequential Organ Failure Assessment (SOFA) Score:
  SOFA score change at Day 3 - baseline, delta = difference between maximum and minimum score during ICU stay, mean/maximum/total daily score during ICU stay, SOFA-3 (score limited to cardiovascular, respiratory and renal function). Measured at baseline and Day 3.
  SOFA score: Minimum possible score is 0, maximum is 24. A higher score meas a worse outcome. Measured at baseline, Day 2 to Day 28.
  SOFA-3 score: Minimum possible score is 0, maximum is 12. A higher score meas a worse outcome. Measured at baseline, Day 2 to Day 28.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
score on a scale
  SOFA change: number analyzed (Participants) | 56 | 56 | 112 | 116
  SOFA change | -0.9 (4.77) | -0.2 (4.87) | -0.5 (4.87) | 0.3 (5.33)
  SOFA Delta score: number analyzed (Participants) | 66 | 70 | 136 | 137
  SOFA Delta score | 4.2 (2.50) | 4.8 (3.80) | 4.5 (3.24) | 3.8 (3.16)
  SOFA maximum score: number analyzed (Participants) | 66 | 70 | 136 | 137
  SOFA maximum score | 10.2 (3.77) | 10.8 (4.46) | 10.5 (4.13) | 9.7 (3.94)
  SOFA mean score: number analyzed (Participants) | 66 | 70 | 136 | 137
  SOFA mean score | 7.957 (3.7546) | 8.319 (3.8129) | 8.143 (3.7751) | 7.644 (3.5105)
  SOFA total score: number analyzed (Participants) | 66 | 70 | 136 | 137
  SOFA total score | 38.9 (33.69) | 54.9 (55.56) | 47.1 (46.78) | 44.1 (48.59)
  SOFA-3 change: number analyzed (Participants) | 64 | 68 | 132 | 152
  SOFA-3 change | -1.7 (2.77) | -0.9 (2.81) | -1.3 (2.80) | -0.9 (2.92)
  SOFA-3 Delta score: number analyzed (Participants) | 66 | 70 | 136 | 137
  SOFA-3 Delta score | 3.5 (1.96) | 3.5 (2.26) | 3.5 (2.11) | 3.1 (2.50)
  SOFA-3 maximum score: number analyzed (Participants) | 66 | 70 | 136 | 137
  SOFA-3 maximum score | 7.2 (2.14) | 7.2 (2.60) | 7.2 (2.38) | 6.8 (2.61)
  SOFA-3 mean score: number analyzed (Participants) | 66 | 70 | 136 | 137
  SOFA-3 mean score | 8.909 (6.5681) | 9.336 (7.2622) | 9.129 (6.9118) | 8.311 (8.0551)
  SOFA-3 total score: number analyzed (Participants) | 66 | 73 | 139 | 139
  SOFA-3 total score | 44.2 (42.36) | 56.4 (51.13) | 50.6 (47.40) | 44.3 (46.45)

16. Secondary Outcome: Change in Renal Function (Creatinine)
Description: Change in renal function as change in creatinine (day 3 - day 1, day 7 - day 1)
Time Frame: day 1, day 3 and day 7
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 70 | 75 | 145 | 151
μmol/L
  creatinine change baseline to day 3: number analyzed (Participants) | 70 | 75 | 145 | 150
  creatinine change baseline to day 3 | -27.9 (85.65) | -11.7 (77.99) | -27.9 (85.65) | -25.6 (109.12)
  creatinine change baseline to day 7 | -46.6 (140.38) | -44.9 (98.44) | -45.7 (120.10) | -50.5 (125.35)

17. Secondary Outcome: Duration of Stay at ICU/ Hospital
Description: Duration of stay at ICU / hospital. The number of participants analyzed differs per row due to missing data.
Time Frame: 90 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
days
  Duration of hospital stay: number analyzed (Participants) | 44 | 42 | 86 | 95
  Duration of hospital stay | 12.3 (11.87) | 13.4 (7.71) | 12.8 (10.2) | 11.2 (7.72)
  Duration of ICU stay: number analyzed (Participants) | 49 | 47 | 149 | 99
  Duration of ICU stay | 9.6 (6.27) | 11.0 (7.26) | 10.3 (6.77) | 9.3 (7.23)

18. Secondary Outcome: Changes of Functional Parameter Mean Arterial Pressure During Stay at ICU
Description: Changes of Mean Arterial Pressure (MAP). Change from baseline to day 28/last day in ICU was calculated (value at day 28 or last collected value minus value at baseline). MAP was collected at screening and daily from day 1 to day 28 or discharge as well as on the follow-up visit day 28. Vital signs were assessed as min/max values within 24 hours except at screening and on the follow-up visit day 28.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
mmHg
  Change from Baseline (minimum) | -7.2 (21.36) | -6.2 (18.44) | -6.7 (19.84) | -6.4 (23.52)
  Change from Baseline (maximum) | 18.9 (23.64) | 17.9 (19.73) | 18.4 (21.64) | 20.2 (21.26)

19. Secondary Outcome: Changes of Functional Parameter Creatinine During Stay at ICU
Description: Changes of creatinine. Measurement for baseline and Day 28 given. Creatinine was measured in the daily blood sample during ICU stay until discharge or Day 28 in a local laboratory assessment.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 71 | 76 | 147 | 152
μmol/L
  Baseline | 189.649 (116.1689) | 199.891 (130.9752) | 194.944 (123.7293) | 192.801 (131.6193)
  Day 28: number analyzed (Participants) | 8 | 12 | 20 | 14
  Day 28 | 84.217 (88.1051) | 79.488 (65.9763) | 81.380 (73.3867) | 153.072 (120.3464)

20. Secondary Outcome: Changes of Functional Parameter Partial Pressure of Oxygen in Arterial Blood(PaO2) / Fraction of Inspired Oxygen (FiO2) During Stay at ICU
Description: Changes of Partial Pressure of Oxygen in Arterial Blood (PaO2) / Fraction of inspired oxygen (FiO2) from baseline to the last observed value are measured. PaO2 and FiO2 was collected if an arterial line was in place. The arterial blood was assessed for PaO2 and FiO2. Both were measured in mmHg.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 65 | 68 | 133 | 136
ratio | 39.83 (155.237) | 63.80 (156.771) | 52.08 (155.896) | 15.91 (164.238)

21. Secondary Outcome: Changes of Functional Parameter Blood Lactate During Stay at ICU
Description: Changes of blood lactate from baseline to Day 28 or discharge. Blood lactate was measured in the daily blood sample from baseline to ICU discharge or until Day 28.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 66 | 70 | 136 | 144
mmol/L | -1.94 (3.133) | -1.54 (5.247) | -1.74 (4.340) | -1.49 (7.158)

22. Secondary Outcome: Changes of Functional Parameter Fluid Balance During Stay at ICU
Description: Changes of fluid balance - Last Observed Value. Percentage of Participants with low (</=1000 mL) and high (>1000 mL) Fluid balance at the last observed value.
  Daily fluid intake will be calculated as the sum of all intravenous and oral fluids. The daily fluid output will be calculated as the sum of the volume of urine output, ultrafiltration fluid, drain fluid, and estimated gastrointestinal losses (including stools only in the presence of profound diarrhea). Insensitive losses will not be taken into account because they are difficult to assess reliably. Daily fluid balance (according to baseline patient weight) will be calculated by subtracting the total fluid output from the total intake.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
percentage of participants
  Low | 80.6 | 84.4 | 82.6 | 80.9
  High | 19.4 | 15.6 | 17.4 | 18.4

23. Secondary Outcome: Changes of Functional Parameter Mid-Regional Pro-Adrenomedullin (MR-proADM) During Stay at ICU
Description: Changes of Mid-Regional pro-Adrenomedullin (MR-proADM) between baseline and last observed value. MR-proADM was measured in the blood samples taken during the ICU stay prior to start of IMP infusion (day 1) and within the time frame of 24 hours (+/- 10 hours) after end of IMP infusion (day 2), at 48 hours, 96 hours and 144 hours after end of infusion (+/- 10 hours) or between scheduled assessments, if discharged earlier from ICU (whatever comes first).
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 61 | 63 | 124 | 127
mmol/L | -5.029 (5.2829) | -4.608 (4.9512) | -4.815 (5.1006) | -4.030 (5.2887)

24. Secondary Outcome: Changes of Functional Parameter Inflammatory Marker Procalcitonine (PCT) During Stay at ICU
Description: Changes of inflammatory marker Procalcitonine (PCT) between baseline and last observed value. PCT was measured in the blood samples taken during the ICU stay prior to start of IMP infusion (day 1) and within the time frame of 24 hours (+/- 10 hours) after end of IMP infusion (day 2), at 48 hours, 96 hours and 144 hours after end of infusion (+/- 10 hours) or between scheduled assessments, if discharged earlier from ICU (whatever comes first).
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 62 | 66 | 128 | 128
ng/mL | -41.402 (125.0852) | -52.661 (78.1064) | -47.208 (103.2929) | -37.219 (78.3425)

25. Secondary Outcome: Changes of Functional Parameter Inflammatory Marker Interleukin-6 (IL-6) During Stay at ICU
Description: Changes of inflammatory marker Interleukin-6 (IL-6) between baseline and last observed value. IL-6 was measured in the blood samples taken during the ICU stay prior to start of IMP infusion (day 1) and within the time frame of 24 hours (+/- 10 hours) after end of IMP infusion (day 2), at 48 hours, 96 hours and 144 hours after end of infusion (+/- 10 hours) or between scheduled assessments, if discharged earlier from ICU (whatever comes first).
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 62 | 66 | 128 | 128
pg/mL | -27648.3 (72859.19) | -37780.4 (119945.41) | -32872.7 (99694.28) | -26236.2 (70315.50)

26. Secondary Outcome: Changes of Functional Parameter Dipeptidyl Peptidase 3 (DPP3) During Stay at ICU
Description: Changes of dipeptidyl peptidase 3 (DPP3) between baseline and last observed value. DPP3 was measured in the blood samples taken during the ICU stay prior to start of IMP infusion (day 1) and within the time frame of 24 hours (+/- 10 hours) after end of IMP infusion (day 2), at 48 hours, 96 hours and 144 hours after end of infusion (+/- 10 hours) or between scheduled assessments, if discharged earlier from ICU (whatever comes first).
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 62 | 66 | 128 | 128
ng/mL | -11.56 (53.030) | -12.47 (42.270) | -12.03 (47.596) | -9.38 (122.031)

27. Secondary Outcome: Vasopressor Use (Drug, Highest Dose)
Description: Vasopressor use (drug, highest dose). Vasopressor use was recorded from admission to ICU at time point of diagnosis of septic shock and daily thereafter from day 1 through day 28 or discharge from ICU (whatever comes first).
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: μg/kg/min
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
μg/kg/min
  OTHER AGENTS FOR LOCAL ORAL TREATMENT: number analyzed (Participants) | 10 | 6 | 16 | 8
  OTHER AGENTS FOR LOCAL ORAL TREATMENT | 1.1236 (1.44760) | 2.1319 (1.53579) | 1.5018 (1.51582) | 1.9888 (2.60114)
  LOCAL HEMOSTATICS: number analyzed (Participants) | 10 | 6 | 16 | 8
  LOCAL HEMOSTATICS | 1.1236 (1.44760) | 2.1319 (1.53579) | 1.5018 (1.51582) | 1.9888 (2.60114)
  ADRENERGIC AND DOPAMINERGIC AGENTS | 3.1414 (7.89069) | 1.7307 (2.03233) | 2.4124 (5.70006) | 1.8276 (4.86110)
  PHOSPHODIESTERASE INHIBITORS: number analyzed (Participants) | 0 | 1 | 1 | 4
  PHOSPHODIESTERASE INHIBITORS |  | 0 (0) | 0 (0) | 3.7763 (1.05962)
  VASOPRESSIN AND ANALOGUES: number analyzed (Participants) | 3 | 2 | 144 | 7
  VASOPRESSIN AND ANALOGUES | 0.0324 (0.02597) | 0 (0) | 0.0289 (0.02265) | 0.0343 (0.02434)
  SYMPATHOMIMETICS, PLAIN: number analyzed (Participants) | 10 | 6 | 16 | 8
  SYMPATHOMIMETICS, PLAIN | 1.1236 (1.44760) | 2.1319 (1.53579) | 1.5018 (1.51582) | 1.9888 (2.60114)
  R03AA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS: number analyzed (Participants) | 10 | 6 | 16 | 8
  R03AA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS | 1.1236 (1.44760) | 2.1319 (1.53579) | 1.5018 (1.51582) | 1.9888 (2.60114)
  R03CA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS: number analyzed (Participants) | 10 | 6 | 16 | 8
  R03CA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS | 1.1236 (1.44760) | 2.1319 (1.53579) | 1.5018 (1.51582) | 1.9888 (2.60114)
  SYMPATHOMIMETICS IN GLAUCOMA THERAPY: number analyzed (Participants) | 10 | 6 | 16 | 8
  SYMPATHOMIMETICS IN GLAUCOMA THERAPY | 1.1236 (1.44760) | 2.1319 (1.53579) | 1.5018 (1.51582) | 1.9888 (2.60114)
  HOMEOPATHIC PREPARATION: number analyzed (Participants) | 10 | 6 | 16 | 8
  HOMEOPATHIC PREPARATION | 1.1236 (1.44760) | 2.1319 (1.53579) | 1.5018 (1.51582) | 1.9888 (2.60114)

28. Secondary Outcome: Patient Reported Outcomes : Quality of Life by Euro-QoL-5
Description: Patient reported outcomes: Quality of Life Form by EuroQoL Group, version "Euro-QoL-5" (day 28 and day 90). Change 1 = Visual analog scale (VAS) at discharge - VAS at day 90. Change 2 = VAS at day 28 - VAS at day 90. Minimum value on the scale is 0, maximum value on the scale is 100. A lower score indicates a worse outcome. As the change between two scores is calculated, a negative number indicates a worsening.
Time Frame: day 28 and day 90
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
score on a scale
  Change 1: number analyzed (Participants) | 27 | 30 | 57 | 71
  Change 1 | -13.4 (22.11) | -19.3 (22.76) | -16.5 (22.45) | -7.6 (27.49)
  Change 2: number analyzed (Participants) | 30 | 33 | 63 | 65
  Change 2 | -11.8 (16.21) | -10.2 (19.40) | -11.0 (17.83) | -5.9 (21.50)

29. Secondary Outcome: Vital Signs
Description: Vital signs: heart rate (beat per minute) Change from baseline to Day 7.
Time Frame: 7 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 40 | 48 | 88 | 80
beats per minute
  Heart Rate Change Day 7 (Maximum) | 5.6 (33.24) | 4.3 (21.85) | 4.9 (27.46) | 13.5 (28.25)
  Heart Rate Change Day 7 (Minimum) | -27.2 (22.91) | -18.5 (20.53) | -22.4 (21.96) | -18.1 (24.49)

30. Secondary Outcome: Penalized Sepsis Support Index (pSSI) at 28 Day Follow-up
Description: Penalized Sepsis Support Index (pSSI) at 28 day follow-up, is a version of the SSI where mortality is given extra weight: Patients being alive duringthe 14 days' follow up will have an SSI ranging up to 14 (as defined above), while patients who died within that period will be assigned a score of "14 plus the number of days not being alive". Thus the weighted SSI score may range between zero and 28. A higher score means a worse outcome.
Time Frame: day 28
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 70 | 75 | 145 | 151
score on a scale | 13.8 (11.34) | 14.8 (10.87) | 14.3 (11.07) | 13.2 (11.36)

31. Secondary Outcome: Vasopressor Use (Drug, Duration)
Description: Vasopressor use (drug, duration). Vasopressor use was recorded from admission to ICU at time point of diagnosis of septic shock and daily thereafter from day 1 through day 28 or discharge from ICU (whatever comes first).
Time Frame: 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 72 | 77 | 149 | 152
days
  OTHER AGENTS FOR LOCAL ORAL TREATMENT: number analyzed (Participants) | 9 | 6 | 15 | 9
  OTHER AGENTS FOR LOCAL ORAL TREATMENT | 1.67 (1.658) | 1.50 (0.837) | 1.60 (1.352) | 1.78 (1.641)
  LOCAL HEMOSTATICS: number analyzed (Participants) | 9 | 6 | 15 | 9
  LOCAL HEMOSTATICS | 1.67 (1.658) | 1.50 (0.837) | 1.60 (1.352) | 1.78 (1.641)
  ADRENERGIC AND DOPAMINERGIC AGENTS: number analyzed (Participants) | 68 | 77 | 145 | 150
  ADRENERGIC AND DOPAMINERGIC AGENTS | 3.00 (1.767) | 3.18 (2.183) | 3.10 (1.994) | 3.34 (2.512)
  PHOSPHODIESTERASE INHIBITORS: number analyzed (Participants) | 0 | 1 | 1 | 3
  PHOSPHODIESTERASE INHIBITORS |  | 0 (0) | 0 (0) | 4.00 (1.732)
  AGENTS FOR TREATMENT OF HEMORRHOIDS AND ANAL FISSURES FOR TOPICAL USE: number analyzed (Participants) | 0 | 0 | 0 | 1
  AGENTS FOR TREATMENT OF HEMORRHOIDS AND ANAL FISSURES FOR TOPICAL USE |  |  |  | 0 (0)
  VASOPRESSIN AND ANALOGUES: number analyzed (Participants) | 4 | 6 | 10 | 11
  VASOPRESSIN AND ANALOGUES | 1.75 (0.500) | 3.00 (1.673) | 2.50 (1.434) | 2.21 (1.701)
  SYMPATHOMIMETICS, PLAIN: number analyzed (Participants) | 9 | 6 | 15 | 10
  SYMPATHOMIMETICS, PLAIN | 1.67 (1.658) | 1.50 (0.837) | 1.60 (1.352) | 1.70 (1.567)
  SYMPATHOMIMETICS, COMBINATIONS EXCL. CORTICOSTEROIDS: number analyzed (Participants) | 1 | 0 | 1 | 1
  SYMPATHOMIMETICS, COMBINATIONS EXCL. CORTICOSTEROIDS | 0 (0) |  | 0 (0) | 0 (0)
  SYMPATHOMIMETICS: number analyzed (Participants) | 1 | 0 | 1 | 1
  SYMPATHOMIMETICS | 0 (0) |  | 0 (0) | 0 (0)
  R03AA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS: number analyzed (Participants) | 9 | 6 | 15 | 9
  R03AA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS | 1.67 (1.658) | 1.50 (0.837) | 1.60 (1.352) | 1.78 (1.641)
  R03CA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS: number analyzed (Participants) | 9 | 6 | 15 | 9
  R03CA ALPHA- AND BETA-ADRENORECEPTOR AGONISTS | 1.67 (1.658) | 1.50 (0.837) | 1.60 (1.352) | 1.78 (1.641)
  SYMPATHOMIMETICS IN GLAUCOMA THERAPY: number analyzed (Participants) | 9 | 6 | 15 | 9
  SYMPATHOMIMETICS IN GLAUCOMA THERAPY | 1.67 (1.658) | 1.50 (0.837) | 1.60 (1.352) | 1.78 (1.641)
  SYMPATHOMIMETICS EXCL. ANTIGLAUCOMA PREPARATIONS: number analyzed (Participants) | 1 | 0 | 1 | 1
  SYMPATHOMIMETICS EXCL. ANTIGLAUCOMA PREPARATIONS | 0 (0) |  | 0 (0) | 0 (0)
  SYMPATHOMIMETICS USED AS DECONGESTANTS: number analyzed (Participants) | 0 | 0 | 0 | 1
  SYMPATHOMIMETICS USED AS DECONGESTANTS |  |  |  | 0 (0)
  HOMEOPATHIC PREPARATION: number analyzed (Participants) | 9 | 6 | 15 | 9
  HOMEOPATHIC PREPARATION | 1.67 (1.658) | 1.50 (0.837) | 1.60 (1.352) | 1.78 (1.641)

32. Secondary Outcome: Change in Renal Function (penKid)
Description: Change in renal function as change in penKid (day 3 - day 1, day 7 - day 1). penKid was measured in the blood samples taken during the ICU stay prior to start of IMP infusion (day 1) and within the time frame of 24 hours (+/- 10 hours) after end of IMP infusion (day 2), at 48 hours, 96 hours and 144 hours after end of infusion (+/- 10 hours) or between scheduled assessments, if discharged earlier from ICU (whatever comes first).
Time Frame: day 1, day 3 and day 7
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 70 | 75 | 145 | 151
pmol/L
  PenKid change baseline to day 3 | -28.3 (57.25) | -21.4 (59.07) | -24.8 (58.10) | -34.8 (63.91)
  PenKid change baseline to day 7: number analyzed (Participants) | 69 | 74 | 143 | 151
  PenKid change baseline to day 7 | -19.5 (83.88) | -19.7 (70.80) | -19.6 (77.11) | -29.8 (83.27)

33. Secondary Outcome: Vital Signs - Blood Pressure
Description: Vital signs: blood pressure - mean arterial pressure (MAP) mmHg Change from baseline to Day 7.
Time Frame: 7 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Arm A | Treatment Arm B | Adrecizumab Overall | Control Group
Number analyzed (Participants) | 40 | 48 | 88 | 80
mmHg
  MAP Change Day 7 (Maximum) | 29.5 (22.26) | 28.2 (16.29) | 28.8 (19.13) | 31.7 (21.09)
  MAP Change Day 7 (Minimum) | -9.6 (17.20) | -6.5 (11.51) | -7.9 (14.37) | -8.7 (18.97)

34. Other Pre Specified Outcome: In Sub-study Key Pharmacokinetic Parameters Peak Plasma Concentrations (Cmax) Are to be Determined in 80 Patients
Description: peak plasma concentrations (Cmax). Time points at which blood samples were taken prior IMP administration, at 30 min, 24 hrs, 48 hrs , 96 hrs, 144 hrs, 648 hrs after IMP administration.
Time Frame: 28 days
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Treatment Arm A | Treatment Arm B
Number analyzed (Participants) | 24 | 29
μg/mL | 38.193 (10.3942) | 86.854 (22.2438)

35. Other Pre Specified Outcome: In Sub-study Key Pharmacokinetic Parameters Time to Cmax (Tmax) Are to be Determined in 80 Patients
Description: Time to Cmax (tmax) in hours (h)
Time Frame: 28 days
Population: Pharmacokinetic Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B
Number analyzed (Participants) | 26 | 30
Participants
  0.25 h | 0 | 1
  0.37 h | 1 | 0
  0.42 h | 2 | 1
  0.45 h | 0 | 1
  0.47 h | 0 | 2
  0.5 h | 17 | 18
  0.57 h | 1 | 0
  0.58 h | 2 | 2
  0.67 h | 1 | 2
  0.73 h | 0 | 1
  2.5 h | 0 | 1
  21.97 h | 0 | 1
  24.75 h | 1 | 0
  25.12 h | 1 | 0

36. Other Pre Specified Outcome: In Sub-study Key Pharmacokinetic Parameter AUC is to be Determined in 80 Patients
Description: systemic exposure : Area under the plasma concentration versus time curve (AUC). Time points at which blood samples were taken prior IMP administration, at 30 min, 24 hrs, 48 hrs , 96 hrs, 144 hrs, 648 hrs after IMP administration.
Time Frame: 28 days
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Treatment Arm A | Treatment Arm B
Number analyzed (Participants) | 10 | 14
h*μg/mL | 4910.33 (1222.414) | 11245.28 (3462.585)

37. Other Pre Specified Outcome: In Sub-study Key Pharmacokinetic Parameter Volume of Distribution is to be Determined in 80 Patients
Description: volume of distribution (V). Time points at which blood samples were taken prior IMP administration, at 30 min, 24 hrs, 48 hrs , 96 hrs, 144 hrs, 648 hrs after IMP administration.
Time Frame: 28 days
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Treatment Arm A | Treatment Arm B
Number analyzed (Participants) | 24 | 29
L | 4.277 (1.9220) | 3.737 (0.9427)

38. Other Pre Specified Outcome: In Sub-study Key Pharmacokinetic Parameter Systemic Clearance is to be Determined in 80 Patients
Description: systemic clearance (CL). Time points at which blood samples were taken prior IMP administration, at 30 min, 24 hrs, 48 hrs , 96 hrs, 144 hrs, 648 hrs after IMP administration.
Time Frame: 28 days
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Treatment Arm A | Treatment Arm B
Number analyzed (Participants) | 10 | 14
L/h | 0.0286 (0.00790) | 0.0280 (0.00826)

39. Other Pre Specified Outcome: In Sub-study Key Pharmacokinetic Parameter Elimination Half-life is to be Determined in 80 Patients
Description: elimination half-life (t½). Time points at which blood samples were taken prior IMP administration, at 30 min, 24 hrs, 48 hrs , 96 hrs, 144 hrs, 648 hrs after IMP administration.
Time Frame: 28 days
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment Arm A | Treatment Arm B
Number analyzed (Participants) | 10 | 14
h | 206.48 (43.809) | 177.90 (44.250)

ADVERSE EVENTS:
Time Frame: All Adverse Events whether serious or non-serious and judged related or unrelated to the study drug occurring during the study period (Day 1 (inclusion and single IMP administration) until 90 days after study drug administration (=Day1)) were collected. The study period was 2 years.
Arm/Group | Treatment Arm A | Treatment Arm B | Control Group
All-Cause Mortality (participants affected / at risk) | 26/72 | 24/77 | 54/152
Serious Adverse Events (participants affected / at risk) | 46/72 | 42/77 | 96/152
Other Adverse Events (participants affected / at risk) | 44/72 | 68/77 | 84/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A (N=72) | Treatment Arm B (N=77) | Control Group (N=152)
Septic shock (Infections and infestations) | 9 (10) | 15 (16) | 26
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Multiple organ dysfunction syndrome (General disorders) | 4 | 7 | 11
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 3 (4)
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 4 (5) | 0 | 1
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 2
Fungal infection (Infections and infestations) | 1 | 0 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Conduction disorder (Cardiac disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 | 1
Urosepsis (Infections and infestations) | 1 (2) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 1 | 1 (2) | 2
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 7
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 2 | 4
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2
Seizure (Nervous system disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 (2) | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 2
Heart valve incompetence (Cardiac disorders) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Weaning failure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 4
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 2 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Embedded device (Product Issues) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Herpes simplex pneumonia (Infections and infestations) | 0 | 1 | 0
Herpes sepsis (Infections and infestations) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Multimorbidity (General disorders) | 0 | 1 | 0
Withdrawal of life support (Surgical and medical procedures) | 0 | 1 | 2
Critical illness (General disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Escherichia peritonitis (Infections and infestations) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 2 (3)
General physical health deterioration (General disorders) | 0 | 1 | 3
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
Osmotic demyelination syndrome (Nervous system disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 2
Endocarditis (Infections and infestations) | 0 | 0 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1
Myocarditis septic (Infections and infestations) | 0 | 0 | 1
Splenic necrosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound abscess (Infections and infestations) | 0 | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 1 (2) | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Primary adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oedema blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A (N=72) | Treatment Arm B (N=77) | Control Group (N=152)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (13) | 10 | 24
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (12) | 14 | 12
Hypernatraemia (Metabolism and nutrition disorders) | 5 | 12 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 6 (7) | 17 (18)
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 8 (9)
Constipation (Gastrointestinal disorders) | 0 | 12 | 7
Cholestasis (Hepatobiliary disorders) | 5 | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT03085758/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03085758/SAP_001.pdf